CLINICAL TRIAL: NCT01651338
Title: Islamic Azad University and Dr Sadre Nabavi Clinic
Brief Title: Quality of Life and Acupuncture on Chronic Pain: A Randomized Study Before and After Performing
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was completed.
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Tahereh Fathi Najafi, ISLAMIC AZAD UNIVERSITY, Islamic Azad University, Sanandaj
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: accupuncture; iaum (Registry Identifier: iaum)
Record Dates: First submitted 2012-07-17; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Pain
Keywords: Acupuncture; quality of life
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- accupuncture, (Experimental): The patients went through acupuncture for 8 -10 sessions and either once or two times a week. The number and the place of needles were 8 -12 for each patient which were located on the right place.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — The patients went through acupuncture for 8 -10 sessions and either once or two times a week. The number and the place of needles were 8 -12 for each patient which were located on the right place.

SUMMARY:
Chronic pains can affect the life quality. This study has performed in the first time in Mashhad.The purpose of the present study was to examine the effect of acupuncture on the life quality of 150 patients who suffered from chronic pain. Some people like performing acupuncture because they believed it's free of risks and beneficial.

In order to achieve this purpose, we had examined the life quality of the patients before and after acupuncture. This study was randomly performed on 150 patients aged between 17-75. They were suffering from chronic pain.

The questionnaire is based on WHO QOL. The questionnaires were filled out once before acupuncture and once 12 weeks after it.

DETAILED DESCRIPTION:
This study was completed on time.

ELIGIBILITY:
Inclusion Criteria:

* aged between 17 - 75 years old,
* suffering from arthritis pains,
* migraine backaches,
* muscular spasms,
* pains in the neck, and in the knee
* duration of disease over 1 year

Exclusion Criteria:

* tacking pain relief
* pregnant women

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
quality of life improvement | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahinfar medical university Fathi Najafi, phD student, Study Director — IAUM
Locations (1):
- Dr sadre Nabavi clinic, Mashhad, Khorasane Razavi, Iran